CLINICAL TRIAL: NCT05826977
Title: CASI-Plus: A Mobile Health (mHealth) Tool for Client Engagement to Improve Ukraine's Assisted Partner Services (APS) Program Workflow and HIV Testing Outcomes (Aim 2)
Brief Title: CASI-Plus mHealth for Ukraine's APS Program (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Public Health Center, Ministry of Health, Ukraine (Unknown)
Responsible Party: Principal Investigator, Nancy Puttkammer, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00015808; 1R21EB032229-01A1 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
Keywords: Ukraine; HIV testing; partner notification
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: In the R21 trial, in one high-volume health facility, researchers will randomize PLWH (N=178) to either the CASI-Plus or standard care (SC) APS workflow, and measure the use of the tool and contact index using routinely-collected data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CASI-Plus (Experimental): The CASI-Plus arm involves use of a tablet-based computerized self-interview tool. This mHealth tool supports the initial assisted partner services (APS) encounter (providing information on how APS works, eliciting names of all sexual or injection partners, screening for risk of intimate partner violence [IPV], and planning for partner notification), and facilitates case management through partner testing (via repeat follow-up surveys to assess for barriers to notification, interest in provider assistance, IPV, and completion of notification).
  Interventions: Behavioral: CASI-Plus
- Standard of care (No Intervention): Standard APS services involve:
  1) Nurses, social workers or doctors introduce APS services to clients during routine health care visits and complete partner elicitation and intimate partner violence (IPV) screening via in-person counseling.
  3) HWs discuss options for partner notification. 4) If index clients opts for a HW to notify the partner, the HW makes multiple contact attempts to contact partners by phone. When index clients return for their regular healthcare services, HW follow up with index clients to check if exposed partners have completed the testing process.
  5) If partners have an unknown HIV status, they are encouraged to complete HIV testing.
  6) Partners who test negative for HIV are referred to HIV prevention services, while those with confirmed HIV diagnoses are linked to HIV care and treatment.

INTERVENTIONS:
Behavioral: CASI-Plus — See arm description
  Arms: CASI-Plus

SUMMARY:
The CASI-Plus mHealth intervention seeks to improve partner elicitation and testing as part of assisted partner services (APS) in Ukraine, through a mHealth client engagement tool using computer-assisted self-interview (CASI). APS is a strategy for contact tracing and HIV testing for the high-risk sexual and needle-sharing partners of patients known to be living with HIV. This implementation science research will provide useful evidence on whether CASI-Plus can improve partner elicitation and HIV testing in a routine APS program operating at scale, toward the ultimate goal of linkage to HIV prevention and treatment services among those at highest risk of HIV. The aim of the study is to assess adoption of CASI-Plus and its impact on contact elicitation in a randomized controlled trial (RCT).

Participants will integrate CASI-Plus as part of the APS services workflow to collect information from clients on sexual partners, needle-sharing partners, and biological children with risk of HIV exposure, and on self-reported partner notification and partner HIV testing outcomes.

The investigators will compare APS clients using CASI-Plus to APS clients receiving standard APS services, to see if the contact index (number of partners named per index client enrolled in APS services) and the HIV testing index (number of partners with unknown HIV status tested per index client enrolled in APS services) increase with use of CASI-Plus.

DETAILED DESCRIPTION:
In December 2016, the World Health Organization (WHO) recommended scale-up of assisted partner notification services (APS) as a strategy to increase HIV testing among persons living with HIV (PLWH). APS offers PLWH assistance to confidentially notify their sex and needle-sharing partners of their exposure and link them to testing and treatment. Randomized controlled trials (RCTs) have shown that APS increases HIV testing and case-finding, and is cost-effective. APS is scalable in routine practice, but typically with lower HIV case-finding than was observed in RCTs. APS outcomes are sub-optimal when recipients only name their current sex partner, or when partner notification and testing does not occur. There are an estimated 240,000 PLWH in Ukraine, of whom roughly three in four know their HIV status. While population-level HIV prevalence is 1.0%, prevalence among persons who inject drugs (PWID) and men who have sex with men (MSM) is 23% and 8%, respectively.

In 2019, the Ukraine Ministry of Health began scaling APS services. Despite trainings that emphasized the need to elicit >1 partner for each index client, health workers (HW) elicited only 1.14 for sexual and needle-sharing partners per index client, on average.16 Only 5.6% of APS clients identified as MSM or PWID and 45.9% of partners with unknown status had not yet completed HIV testing after 30 days.

The CASI-Plus mHealth intervention seeks to improve partner elicitation and testing, through a mHealth client engagement tool using computer-assisted self-interview (CASI). The CASI-Plus tool supports the initial APS encounter (providing information on how APS works, eliciting names of all sexual or injection partners, screening for risk of intimate partner violence [IPV], and planning for partner notification), and facilitates case management through partner testing (via repeat follow-up surveys to assess for barriers to notification, interest in provider assistance, IPV, and completion of notification). While CASI has reduced social desirability bias in surveys of sexual behavior across diverse settings, it has not yet been used in APS programs in low- or middle-income countries (LMICs). This implementation science research will provide useful evidence on whether CASI-Plus can improve partner elicitation and HIV testing in a routine APS program operating at scale, toward the ultimate goal of linkage to HIV prevention and treatment services among those at highest risk of HIV.

Aim 1 (R21): Conduct formative research from health worker and client perspectives to design the CASI-Plus mHealth intervention. Approach: The investigators will complete in-depth interviews with APS clients (N=10) and focus group discussions with HWs (N=2 groups of 8 HWs) to elicit barriers to partner elicitation and testing, use this information to design the CASI-Plus tool and its integration within the APS workflow, and test the tool for technical performance, usability, and acceptability. Hypothesis: CASI-Plus will be perceived by both clients and HWs as easy to navigate, acceptable, and technically sound. [NOTE: Aim 1 is covered under a separate submission to ClinicalTrials.gov]

Aim 2 (R21): In a RCT, assess adoption of CASI-Plus and its impact on contact elicitation. Approach: In one high-volume health facility, the investigators will randomize PLWH (N=154) to either the CASI-Plus or standard care (SC) APS workflow, and measure the use of the tool and contact index using routinely-collected data. Hypothesis: Clients will complete initial and follow-up surveys, and will report more partners when using the tool.

The proposed research team brings together experienced researchers, APS program specialists, and digital health specialists from the University of Washington (UW) and the Ministry of Health's Public Health Center (PHC). The project builds upon the existing national platform for APS within public-sector HIV clinics, and lays the foundation for a simple intervention to optimize APS delivery which could be evaluated for implementation outcomes and effectiveness at scale in a future cluster-randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria for APS Index Clients (R21 Aim 2)

1. consent to participate in APS services and the study;
2. are 18 years or older;
3. have been diagnosed with HIV and enrolled in care;
4. have not previously participated in APS services at another health facility; and
5. have access to a personal cell phone and internet.

Exclusion Criteria Does not meet one or more inclusion criteria

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Contact index | Baseline measurement
  This is the primary outcome for the R21 study, measured during the initial APS encounter, at client enrollment into the study. Number of partners named per index client. This outcome will be measured through routine APS program data sources including APS case files and the HIV management information system (MIS) electronic health record system.
Testing index | Measured at 8 weeks
  This is a secondary outcome for the Aim 2 Study. Number of partners with unknown HIV status tested per index client. This outcome will be measured through routine APS program data sources including APS case files and the HIV MIS electronic health record system.

SECONDARY OUTCOMES:
CASI-Plus tool system usability | Measured at study completion, on average after 8-12 weeks
  System Usability Scale (Bangor, 2008). This is a 10-item instrument with 5-point Likert scale response options, such as "I found the tool unnecessarily complex" or "I would imagine that most people would learn to use this tool very quickly".
Adoption of CASI-Plus | Measured between baseline and 8 weeks
  Percentage of clients responding to >=1 follow-up survey, based on CASI-Plus paradata and APS case files
Level of engagement with CASI-Plus | Measured between baseline and 8 weeks
  Average number of direct engagements between index clients and HW through case closure, based on CASI-Plus paradata and APS case files

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Puttkammer, PhD, MPH, Principal Investigator — University of Washington
Locations (2):
- Ukraine (2):
  - • Municipal Enterprise "Chernihiv Regional Hospital" of the Chernihiv Regional Council "Center for HIV/AIDS and Hepatitis Prevention", Chernihiv, Chernihiv Oblast
  - • Municipal Enterprise "Dnipropetrovsk Regional Medical Center for Socially Significant Diseases" of the Dnipropetrovsk Regional Council, Dnipro, Dnipro

IPD SHARING:
Plan to Share IPD: Yes
Shared individual participant data (IPD) will include IPD that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices). Anyone who wishes to access the data and who provides a methodologically sound proposal, may request access IPD. Researchers will be asked to submit a request in writing describing their qualifications including their certification by their local institutional review board (IRB), analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data. They will be required to agree in writing that they will not share the data with others, will use it only for the research purpose(s) delineated, and will return or destroy the data upon completion. Proposals should be directed to Nancy Puttkammer (nputt@uw.edu). Given the sensitive nature of the data we are collecting, including HIV diagnosis, the data will not be shared in a public access file.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The HIV MIS and APS register data are considered to be owned by the Ukraine Ministry of Health's Public Health Center (PHC). The Principal Investigator (PI) will share the secondary data obtained for the study from PHC's routine data systems with other researchers, upon written documentation of PHC agreement.